CLINICAL TRIAL: NCT02528851
Title: Cardiorespiratory Effects of "Higher" Versus "Equivalent" CPAP Upon Extubation From High Endotracheal Airway Pressures in Preterm Infants: A Randomized Cross-Over Trial
Brief Title: Cardiorespiratory Effects of "Higher" Versus "Equivalent" CPAP Upon Extubation From High EAP in Preterm Infants
Acronym: CO-PAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Souvik Mitra, MD, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-PAP
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Preterm Infant
Keywords: CPAP; preterm; cardiac output
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher CPAP (Experimental): Infants extubated to CPAP level 2cm H2O higher than extubation EAP
  Interventions: Procedure: Extubation from endotracheal mechanical ventilation to CPAP
- Equivalent CPAP (Active Comparator): Infants extubated to CPAP equivalent to extubation EAP
  Interventions: Procedure: Extubation from endotracheal mechanical ventilation to CPAP

INTERVENTIONS:
Procedure: Extubation from endotracheal mechanical ventilation to CPAP — Following randomization, the infants will be extubated to the "higher" CPAP group (CPAP level 2cm H2O higher than extubation EAP) or "equivalent" CPAP group (CPAP level equal to the extubation EAP) based on their allocation.

SUMMARY:
The aim of this study is to compare the cardiovascular and respiratory effects of "higher" versus "equivalent" CPAP pressures post-extubation from high endotracheal airway pressures (EAP), defined as at least 8 cm H2O (water), in the form of a randomized controlled cross-over trial. Endotracheal airway pressure (EAP) will be defined as mean airway pressure (MAP) [if on high frequency ventilation] or positive end-expiratory pressure (PEEP) [if on conventional ventilation] at time of extubation. Participants will be randomized to "higher" CPAP group (CPAP level 2cm H2O higher than the extubation EAP) or "equivalent" CPAP group (CPAP level equal to the extubation EAP) before undergoing crossover to the other arm. We hypothesize that "higher" CPAP levels, when compared to "equivalent" CPAP levels, do not adversely impact the cardiorespiratory status when a patient is extubated from high EAP.

DETAILED DESCRIPTION:
Extubation readiness of the enrolled infants will be determined solely by and at the discretion of the medical team. All enrolled infants will be checked to re-confirm eligibility prior to extubation. Those enrolled infants who are ventilated on EMV (endotracheal mechanical ventilation) with an airway pressure of 8-11 cm H2O at the time when they are deemed extubation-ready by the team will be eligible for randomization. Once eligibility for randomization is assessed, the study coordinator will notify the research team who will immediately perform a bedside functional echocardiography to assess cardiac output and PDA (patent ductus arteriosus) status. In addition, the lung compliance (as measured by the ventilator) will be recorded. If a PDA exists and is found to be hemodynamically significant, then the infant meets one of the exclusion criteria and will be ineligible for randomization.

Once eligibility is confirmed, infants will be randomized using sequentially numbered sealed opaque envelopes. The sequence of the randomization will be pre-determined using a computer generated algorithm, and sealed envelopes will be created by study coordinator. Once randomized, the infants will be extubated to the "higher" CPAP group (CPAP level 2cm H2O higher than extubation EAP) or "equivalent" CPAP group (CPAP level equal to the extubation EAP) based on their allocation.

After ensuring that the infants are stable for one hour (based on pre-defined clinical instability criteria) cardiac output will be measured using bedside functional echocardiography by members of the research team blinded to the allocation. To ensure blinding the research coordinator will cover the relevant digital display of the ventilator/CPAP machine (with opaque craft paper and tape) immediately prior to the echocardiography. Other aforementioned outcomes will be recorded by the blinded investigator using standardized data collection forms. Once all outcome data are collected, the infants will cross-over to the opposite arm of the trial and a similar assessment protocol will be followed after one hour. The study protocol will be considered completed when the second set of measurements is obtained and further respiratory management will be guided by the medical team.

SAFETY ASSURANCE At any point during the study, emergence of any one of the clinical instability criteria will prompt the nursing staff to notify the medical team who would immediately assess the infant. If the infant shows signs of clinical instability the medical team will evaluate the infants' clinical condition as per a pre-defined checklist. When all the troubleshooting points mentioned in the checklist are addressed by the medical team and the infant is deemed clinically unstable, the infant would be immediately removed from the study protocol and parents of the subject will be notified. To ensure that no other factor affects the hemodynamic status of the infants during the study, the total fluid intake would remain the same and no caffeine citrate would be administered during the period of pre and post extubation assessment of cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants less than 37 weeks of gestation who are mechanically ventilated with Endotracheal Airway Pressure (EAP) ≥ 8 cm H2O at time of extubation as per the medical team.

Note: The decision to extubate a subject, and EAP at time of extubation, will solely be that of the medical team, and is in no way dictated by the study protocol.

Exclusion Criteria:

* Infants on EMV with EAP> 11 cmH2O at the time of extubation
* Congenital or acquired abnormality of upper airway
* Major gastrointestinal disorder or complication
* Suspected/proven chromosomal/genetic abnormality
* Suspected/confirmed sepsis being treated at time of extubation
* Unresolved hemodynamically significant patent ductus arteriosus (with or without inotropic support) at time of extubation
* Congenital structural heart diseases
* Infants requiring vasopressor and/or inotropic support at time of extubation
* Persistent pulmonary hypertension requiring treatment with vasopressors/inhaled nitric oxide/sildenafil at time of extubation
* Any unplanned extubation in infants otherwise meeting the inclusion criteria.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular output | One hour after each intervention
  We will use the formula LVO = [LV Outflow Tract (LVOT) area x Quantity of blood across LVOT x heart rate]/body weight (ml/kg/min). The details of measurement of each component of the equation are as follows:
  * LVOT area = π (LV outflow tract diameter/2)2. LV outflow tract diameter will be measured in the parasternal long axis in late systole immediately distal to the valve orifice using the leading edge technique.
  * Quantity of blood across the LVOT: To be measured using the VTI (velocity time integral) from pulsed Doppler echocardiography from the modified apical view (5-chamber view)

SECONDARY OUTCOMES:
Heart rate | One hour after each intervention
Blood pressure | One hour after each intervention
  non-invasive cuff blood pressure
abdominal wall girth | One hour after each intervention
  measured using a tape measure at the level of the umbilicus
Silverman-Andersen respiratory score | One hour after each intervention
Lung compliance | Pre-extubation measurement in all recruited infants
  Dynamic compliance would be noted from the ventilator control panel (defined as change in volume per unit change in pressure)
Inferior vena caval diameter | One hour after each intervention
  Using functional echocardiography mean inferior vena caval diameter will be measured. Mean inferior vena cava diameter (IVCD), expressed as[(IVCD in inspiration + IVCD in expiration)/2]
Superior vena caval flow | One hour after each intervention
  We will use the formula SVC flow = [Mean SVC area x Quantity of blood across SVC x heart rate]/body weight (ml/kg/min).
  * Mean SVC area = π (Mean SVC diameter /2)2. Mean SVC diameter will be measured in the parasternal long axis with the beam in a true sagittal plane and angled to the right of the ascending aorta. The mean of the maximum and minimum internal diameters will be taken for flow measurement to account for the variation in vessel diameter during the cardiac cycle.
  * Quantity of blood across the SVC: To be measured using the VTI (velocity time integral) from pulsed Doppler echocardiography from a low subcostal view

CONTACTS AND LOCATIONS:
Overall Officials: Souvik Mitra, MD, Principal Investigator — McMaster University